CLINICAL TRIAL: NCT01230918
Title: Technetium-NC100692 SCintigraphy to Detect avB3 Integrin Expression as a mARker of Fibrosis in Hypertrophic Cardiomyopathy and Acute Coronary Syndrome: the SCAR Study
Brief Title: Study to Develop a Non-invasive Marker for Monitoring Myocardial Fibrosis
Acronym: SCAR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Costs of study procedures has changed and escalated and became prohibitive.
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Terrence Ruddy, Principal Investigator, Ottawa Heart Institute Research Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HI Protocol #2009641-01H
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Hypertrophic Cardiomyopathy; Acute Coronary Syndrome
Keywords: Hypertrophic Cardiomyopathy; Acute Coronary Syndrome; Myocardial Fibrosis; Fibrogenesis; Intimal Hyperplasia; Sudden Death; avB3 Integrin Expression
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Acute Coronary Syndrome; Death, Sudden | interventions — technetium 99m NC 100692

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic Imaging (Experimental): A single dose of 800 to 1100 mBq of 99mTc-NC100692 radiopharmaceutical will be injected. Serial cardiac nuclear imaging will be done over a 3 hour period.
  Interventions: Radiation: 99mTc-NC100692

INTERVENTIONS:
Radiation: 99mTc-NC100692 — HCM and ACS subjects: 99mTc-NC100692 SPECT scan, CMR and echocardiography images will be obtained and compared.
  Normal control: 99mTc-NC100692 SPECT scan, CMR and echocardiography imaging obtained for comparison with HCM and ACS images.

SUMMARY:
The objective is to determine whether 99Technetium-NC100692 uptake in patients with ACS (MI) can serve as a marker for scar formation as detected by contrast-enhanced MRI during the process of myocardial remodelling after the ischemic insult.

Comparison of ACS and HCM Populations:

The primary objective is to determine whether TcNC100692 imaging is able to quantify the extent to which myocardial fibrogenesis occurring early post myocardial infarction differs from that in patients with hypertrophic cardiomyopathy.

The primary hypothesis is that since fibrogenesis is known to occur most intensely in the first days to weeks post myocardial infarction, while it is a more protracted, less predictable process in HCM, there will be significantly more TcNC100692 uptake in the early post-ACS population than in the HCM population.

Control Population:

Normal control images will allow for differentiation of uptake in the myocardium.

DETAILED DESCRIPTION:
HCM Population:

The primary objective is to determine whether fibrosis detected by MRI and 99mTc-NC100692 uptake in patients with HCM are associated. The secondary objective is to determine whether 99mTc-NC100692 uptake correlates on a segmental basis with fibrosis visualised by late Gd-enhancement MRI. The tertiary objective is to evaluate the relationship between the extent of fibrosis assessed by 99mTc-NC100692 uptake and mean longitudinal strain as determined by speckle tracking echocardiography.

The primary hypothesis is that there is an increased uptake of 99mTc-NC100692 in patients with HCM fibrosis detected by MRI. The secondary hypothesis is that the location and extent of increased 99mTc-NC100692 uptake will correlate with localization and extent measurements of fibrosis by Gd-enhanced magnetic resonance imaging. The tertiary hypothesis is that the extent of fibrosis assessed by the number of segments with and the magnitude of 99mTc NC100692 uptake will correlate with mean longitudinal strain as determined by speckle tracking echocardiography.

ACS Population:

The objective is to determine whether 99Technetium-NC100692 uptake in patients with ACS (MI) can serve as a marker for scar formation as detected by contrast-enhanced MRI during the process of myocardial remodelling after the ischemic insult.

The primary hypothesis is that there is an increased uptake of 99Technetium-NC100692 in patients following an ACS event (MI) and that the location and extent of increased 99Technetium-NC100692 uptake will correlate with the presence and extent of scar as detected by contrast-enhanced magnetic resonance imaging.

Normal Control Population:

Preliminary analysis of images from HCM population showed a diffuse, low grade uptake of 99Technetium-NC100692 in non-hypertrophied myocardial segments. Although not entirely unexpected, comparison with control images will allow for quantification of low grade fibrosis and low grade uptake.

ELIGIBILITY:
HCM Population:

Inclusion Criteria:

* Diagnosis of HCM as defined as: Interventricular septal thickness greater than 12 mm on a 2D echocardiogram, or septal: posterior wall thickness as measured on parasternal long axis view of >1.3 in the absence of secondary causes of cardiac hypertrophy such as aortic stenosis and systemic hypertension.

Exclusion Criteria:

* Concomitant diseases that can lead to myocardial hypertrophy including valvular heart disease and uncontrolled hypertension. If HCM is proven by either the presence of a family history of HCM or through genotyping, patients with controlled hypertension will not be excluded.
* Documented coronary artery disease including a history of previous myocardial infarction or coronary intervention or revascularization.
* Known diabetic cardiomyopathy.

ACS Population:

Inclusion Criteria:

* Diagnosis of ACS, either NSTEMI as determined by positive myocardial markers or STEMI patients who have an onset of symptoms 12 hours or less before presentation and an ST-segment elevation of at least 1 mm in two or more contiguous limb leads or of at least 2 mm in two or more contiguous precordial leads during prehospital 12-lead ECGs. Patients will undergo 99mTc-NC100692 imaging within 1 week of acute myocardial infarction.

Exclusion Criteria:

* Patients presenting with an acute STEMI secondary to an occlusive thrombus who were revascularized with coronary artery bypass surgery.
* Patients with a known prior history of cardiomyopathy of any cause (ex. ischemic, hypertrophic, infiltrative, idiopathic dilated), preceding the index referral for primary PCI.
* Hemodynamic instability or cardiogenic shock.

Normal Control:

Inclusion Criteria:

* No clinically significant chronic or acute illness as determined by history, echocardiogram and/or available reports.

Exclusion Criteria:

* Subjects with pre-existing confounding factors, such as hypertension, diabetes mellitus, hyperlipidemia, CAD, known structural heart disease, left ventricular dysfunction, previous cerebrovascular event, malignancy, connective tissue or inflammatory disease, chronic infection, and hepatic or renal impairment will be excluded.
* Possess abnormal cardiac structure and function after examination with ECHO

All populations:

Inclusion Criteria:

* The subject is greater than or equal to 18 years of age at study entry.
* Before any study procedure is carried out, the subject is able and willing to comply with study procedures and has provided signed and dated informed consent, including permission to access medical records.
* The subject is male, or a female who is either surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy), postmenopausal (cessation of menses for more than 1 year), non-lactating, or of childbearing potential for whom the result of a urine pregnancy test performed before administration of IMP is negative.

Exclusion Criteria:

* Hypersensitivity to any component of 99mTc-NC100692 injection (e.g. p- aminobenzoate).
* Pregnancy.
* Unwillingness to provide and sign for informed consent.
* Creatinine clearance <30 ml/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-05; Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
TcNC100692 uptake | 3 hours
  The primary objective is to determine whether TcNC100692 imaging is able to quantify the extent to which myocardial fibrogenesis occurring early post myocardial infarction differs from that in patients with hypertrophic cardiomyopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Terrence Ruddy, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada